CLINICAL TRIAL: NCT07004075
Title: An Open-label, Randomized, Multi-center Phase III Clinical Study: Aim to Evaluate the Efficacy and Safety of FCN-159 Monotherapy Versus the Treatment by Investigator's Choice in Patients With Pediatric Low-grade Glioma Harboring KIAA1549-BRAF Fusion or BRAF V600E Mutation
Brief Title: FCN-159 Monotherapy Versus Chemotherapy by Investigator's Choice in Pediatric Low-grade Glioma Patients With BRAF Alteration
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCN-159-010
Record Dates: First submitted 2025-06-03; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Low-grade Glioma; Pediatric Low-grade Gliomas; pLGG With BRAF Alteration
MeSH Terms: interventions — Vindesine; Carboplatin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: Luvometinib (Experimental): FCN-159, 5 mg/m^2, once daily, continuous oral administration
  Interventions: Drug: Luvometinib
- Comparator: investigator's choice of chemotherapy (Active Comparator): Chemotherapeutic Agent COG-V/C, intravenous solution for injection Carboplatin + Vindesine, intravenous solution for injection Carboplatin, intravenous solution for injection Temozolomide, orally Day 1 to Day 5 of each 28 days as a cycle
  Interventions: Biological: Chemotherapeutic Agent COG-V/C Carboplatin + Vindesine, Carboplatin, Temozolomide

INTERVENTIONS:
Drug: Luvometinib — Luvometinib oral tablet
  Arms: Experimental arm: Luvometinib
Biological: Chemotherapeutic Agent COG-V/C Carboplatin + Vindesine, Carboplatin, Temozolomide — Investigator's choice of chemotherapy administered IV or orally
  Arms: Comparator: investigator's choice of chemotherapy

SUMMARY:
An open-label, randomized, multi-center phase III clinical study: Aim to evaluate the efficacy and safety of FCN-159 monotherapy versus the treatment by investigator's choice in patients with pediatric low-grade glioma harboring KIAA1549-BRAF fusion or BRAF V600E mutation

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients aged between ≥ 2 years and < 18 years; regardless of male or female.
2. Histologically and/or cytologically confirmed diagnosis of low-grade glioma (pLGG diagnosis as Grade 1 or 2 according to the 2021 WHO classification of CNS).
3. KIAA1549-BRAF fusion or BRAF V600E mutation-positive.
4. Patients requiring systemic therapy as determined by the investigator, including patients having disease recurrence or progression, or residual disease of surgery, or unresectable.
5. At least one intracranial measurable lesion that can be reproducibly measured in two dimensions on T2-FLAIR, with the minimum size of the bi-perpendicular diameter of ≥ 10 mm, and can be visible on two or more imaging slice.

6. Karnofsky performance score or Lansky performance score ≥ 70. 7．Adequate organ function within 14 days before enrollment.

Exclusion Criteria:

1. Patients who have previously received any of the following treatments:

   1. Patients who have received chemotherapy drugs or traditional Chinese medicines or herbals with definitive anti-tumor treatment within 4 weeks preceding the first dose of investigational drug;
   2. Patients who have received growth factors that promote platelet or leukocyte count or function within 14 days preceding the first dose of investigational drug;
   3. Patients who received radiotherapy, surgery or immunotherapy within 4 weeks preceding the first dose of investigational drug;
   4. Patients who have participated in other interventional clinical trials within 4 weeks before receiving the first dose of investigational drug;
   5. Patients who have received live vaccines within 4 weeks preceding the first dose of investigational drug, or patients who have received inactivated vaccines and mRNA vaccines within 14 days preceding the study treatment;
   6. Patients who have previously received any other MEK 1/2 inhibitors such as Selumetinib or BRAF inhibitors such as Dabrafenib.
2. Patients with high-grade gliomas, as well as schwannoma, subependymal giant cell astrocytoma (tuberous sclerosis), and diffuse intrinsic pontine gliomas (even if the histological diagnosis is WHO Grade 1 or 2).
3. Patients who require endotracheal intubation for assisted ventilation or tracheotomy should be excluded.
4. Patients who have uncontrollable epilepsy as assessed by the investigator.
5. Patients with dysphagia, active GI diseases, malabsorption syndrome, or other conditions that will interfere with the absorption of the investigational drug.
6. Patients with clinically significant active bacterial, fungal or viral infections, including hepatitis B virus surface antigen positive and hepatitis B virus DNA exceeding 1000 IU/ml. Hepatitis B carriers are allowed to be enrolled. Patients with positive hepatitis C virus (HCV) antibody test; those who have confirmed human immunodeficiency virus (HIV) infection, and are unwilling to undergo HIV testing.
7. Patients with history or current evidence of retinal vein obstruction (RVO), retinal pigment epithelial detachment (RPED), central retinal vein occlusion, glaucoma, and other significant abnormalities in ophthalmological examinations.
8. Interstitial pneumonia, including clinically significant radiation pneumonitis.
9. Grade 3 creatine phosphokinase increased (>5 × ULN - 10 × ULN).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Compare the progression free survival (PFS) of FCN-159 versus chemotherapy by IRC | up to 48 months
  PFS assessed per RANO-LGG criteria by IRC, and defined as the time from randomization to the first recorded progressive disease or death from any cause, whichever is first

SECONDARY OUTCOMES:
PFS of FCN-159 versus chemotherapy by INV | up to 48 months
  PFS assessed per RANO-LGG criteria by inverstigator
Objective response rate (ORR) of FCN-159 versus chemotherapy | up to 48 months
  ORR assessed per RANO-LGG criteria,and defined as the proportion of patients with confirmed complete response (CR), partial response (PR) or minor response (MR)
Clinical benefit rate (CBR) of FCN-159 versus chemotherapy | up to 48 months
  CBR is defined as the proportion of patients with confirmed CR, PR, MR and SD lasting ≥24 weeks as assessed based on the RANO-LGG criteria
Duration of overall response (DOR) of FCN-159 versus chemotherapy | up to 48 months
  DOR is defined as the time from the date of the first CR, PR or MR to the first recorded tumor progression or death (death due to any cause), whichever occurs earlier
Time to response (TTR) of FCN-159 versus chemotherapy | up to 48 months
  TTR is defined as the time from the first dose of the investigational drug to the first confirmed CR, PR or MR based on the RANO-LGG criteria
Overall survival (OS) of FCN-159 vesus chemotherapy | up to 48 months
  OS is defined as the time from the first dose of the investigational drug to death by any cause
Safety of FCN-159 versus chemotherapy | up to 48 months
  Number of Participants With Adverse Events (AEs) of treated participants

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China